CLINICAL TRIAL: NCT00389909
Title: Evaluation of Dosing Chart Taking Into Account Age and Gender for Calculating the First Dose of Doxapram in Premature Infants
Brief Title: Dosing Chart for Calculating the First Dose of Doxapram in Premature Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jean Michel Hascoet (Other)
Responsible Party: Sponsor-Investigator, Jean Michel Hascoet, Professor, Maternite Regionale Universitaire
Organization: Maternite Regionale Universitaire (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRAP060309
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Premature Infants; Apnea
Keywords: Premature infants; Apnea; Doxapram; pharmacokinetics
MeSH Terms: conditions — Premature Birth; Apnea | interventions — Doxapram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Treatment based on patient weight;
  Interventions: Drug: Doxapram
- 2 (Active Comparator): Treatment based on a chart taking into account weight, age and gender
  Interventions: Drug: Doxapram

INTERVENTIONS:
Drug: Doxapram — Dosing comparison between fixed scheduled and sex related dosage.
  Dosing related to weight only versus chart taking into account weight, age and gender.
  Other Names: Dopram

SUMMARY:
Doxapram is used to stimulate respiration. For a given dose, the fluctuations in concentrations observed in infants' blood may be wide, leading to a risk of lack of efficacy or of toxic effects. Two factors are linked to these fluctuations: age and gender. The aim of this study is to compare a dosage regimen based only on patient's weight, to another one using a dosing chart taking into account weight, age and gender.

DETAILED DESCRIPTION:
Doxapram is a drug used to stimulate respiration in neonates prematurely born and failing to breathe. For a given dose, the fluctuations in concentrations of drug observed in infants' blood might be wide, leading to a risk of lack of efficacy of the treatment or of toxic effects. Two factors are linked to these fluctuations: age and gender. The aim of our study is to compare a dosage regimen based only on patient's weight, and another one using a dosing chart taking into account not only weight but also age and gender to prescribe the initial dose of doxapram. The final goal of this trial is to improve efficacy and tolerance of doxapram by minimizing the fluctuations in blood drug levels in premature neonates.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants (<37 weeks gestation)
* More than 1 significant Apnea q 8h (> 20 sec or < 20 sec with bradycardia or desaturation)
* Already treated with caffeine

Exclusion Criteria:

* Intubation
* congenital malformation
* symptomatic apnea

Ages: 1 Week to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2006-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Plasma level of Doxapram and its active metabolite (ketodoxapram) at 48 hours after the onset of treatment. | 48 Hours

SECONDARY OUTCOMES:
Efficacy (rate of significant apnea) | 1 Week

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Jeanne BOUTROY, PhD, Study Director — INSERM, France; Jean-Michel HASCOET, MD, Principal Investigator — University of NANCY France
Locations (2):
- France (2):
  - Maternite Regionale Universitaire, Nancy
  - Hopital des Enfants, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbe F, Hansen C, Badonnel Y, Legagneur H, Vert P, Boutroy MJ. Severe side effects and drug plasma concentrations in preterm infants treated with doxapram. Ther Drug Monit. 1999 Oct;21(5):547-52. doi: 10.1097/00007691-199910000-00011. PMID 10519454
- [Derived] Greze E, Benard M, Hamon I, Casper C, Haddad FE, Boutroy MJ, Hascoet JM. Doxapram Dosing for Apnea of Prematurity Based on Postmenstrual Age and Gender: A Randomized Controlled Trial. Paediatr Drugs. 2016 Dec;18(6):443-449. doi: 10.1007/s40272-016-0192-2. PMID 27612991